CLINICAL TRIAL: NCT00490035
Title: A Multi-center, Double-blind, Parallel-group, Placebo Controlled, Randomized Study: Evaluation of the Efficacy and Safety of Brivaracetam in Subjects (>= 16 to 70 Years Old) With Partial Onset Seizures.
Brief Title: Double-blind, Randomized Study Evaluating the Efficacy and Safety of Brivaracetam in Adults With Partial Onset Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma SA (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N01252; 2006-006344-59 (EudraCT Number)
Record Dates: First submitted 2007-06-21; First posted 2007-06-22 (Estimated); Results first posted 2016-04-13 (Estimated); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Epilepsy
Keywords: Epilepsy; Brivaracetam; Partial Onset Seizures
MeSH Terms: conditions — Epilepsy | interventions — brivaracetam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Matching Placebo tablets administered twice a day
  Interventions: Other: Placebo
- Brivaracetam 20 mg/day (Experimental): Brivaracetam 20 mg/day, 10 mg administered twice a day
  Interventions: Drug: Brivaracetam
- Brivaracetam 50 mg/day (Experimental): Brivaracetam 50 mg/day, 25 mg administered twice a day
  Interventions: Drug: Brivaracetam
- Brivaracetam 100 mg/day (Experimental): Brivaracetam 100 mg/day, 50 mg administered twice a day
  Interventions: Drug: Brivaracetam

INTERVENTIONS:
Other: Placebo — Daily oral dose of two equal intakes, morning and evening, of Placebo in a double-blinded way for the 12-week Treatment Period
  Arms: Placebo
Drug: Brivaracetam — Daily oral dose of two equal intakes, morning and evening, of Brivaracetam 20 mg /day in a double-blinded way for the 12-week Treatment Period
  Arms: Brivaracetam 20 mg/day
Drug: Brivaracetam — Daily oral dose of two equal intakes, morning and evening, of Brivaracetam 50 mg /day in a double-blinded way for the 12-week Treatment Period.
  Arms: Brivaracetam 50 mg/day
Drug: Brivaracetam — Daily oral dose of two equal intakes, morning and evening, of Brivaracetam 100 mg /day in a double-blinded way for the 12-week Treatment Period.
  Arms: Brivaracetam 100 mg/day

SUMMARY:
This study will evaluate the efficacy and safety of Brivaracetam to support the submission file in the indication of adjunctive treatment in adolescents and adults with partial onset seizures.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were from 16 to 70 years, both inclusive. Subjects under 18 years of age were only included where legally permitted and ethically accepted
* Subjects with well-characterized focal epilepsy or epileptic syndrome according to the International League Against Epilepsy (ILAE) classification
* Subjects had a history of partial onset seizures (POS) whether or not secondarily generalized (Type I seizures according to the ILAE classification)
* Subjects had at least 2 POS whether or not secondarily generalized per month during the 3 months preceding Visit 1
* Subjects had at least 8 POS whether or not secondarily generalized during the 8-Week Baseline Period
* Subjects were uncontrolled while treated by 1 to 2 permitted concomitant antiepileptic drugs (AEDs). Vagal nerve stimulation was allowed and was not counted as a concomitant AED

Exclusion Criteria:

* History or presence of seizures occurring only in clusters (too frequently or indistinctly separated to be reliably counted) before Visit 3
* History or presence of status epilepticus during the year preceding Visit 1 or during Baseline

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2007-09; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (76):
- Belgium (4):
  - 13, Ghent
  - 19, La Louvière
  - 12, Liège
  - 10, Sankt Vith
- Finland (4):
  - 44, Kuopio
  - 41, Oulu
  - 42, Seinäjoki
  - 43, Tampere
- France (11):
  - 60, Angers
  - 56, Béthune
  - 62, Bron
  - 57, Dijon
  - 53, Lille
  - 52, Montpellier
  - 64, Nancy
  - 54, Paris
  - 51, Rennes
  - 61, Roanne
  - 55, Strasbourg
- Germany (10):
  - 76, Bad Berka
  - 73, Berlin
  - 79, Bernau
  - 78, Bielefeld
  - 74, Freiburg im Breisgau
  - 75, Kehl-Kork
  - 77, Mainz
  - 70, München
  - 72, Radeberg
  - 71, Ulm
- Hungary (3):
  - 94, Budapest
  - 90, Debrecen
  - 92, Pécs
- India (9):
  - 256, Bangalore
  - 257, Bangalore
  - 253, Hyderabad
  - 258, Jaipur
  - 255, Kolkata
  - 250, Lucknow
  - 259, Mumbai
  - 270, Pune
  - 251, Pune Maharashtra
- Italy (5):
  - 104, Bologna
  - 105, Foggia
  - 101, Perugia
  - 103, Roma
  - 107, Roma
- Netherlands (3):
  - 124, Breda
  - 125, The Hague
  - 122, Zwolle
- Poland (14):
  - 142, Bialystok
  - 143, Gdansk
  - 153, Grodzisk Mazowiecki
  - 147, Katowice
  - 151, Katowice
  - 141, Kielce
  - 150, Krakow
  - 148, Lodz
  - 144, Lublin
  - 152, Poznan
  - 146, Szczecin
  - 140, Warsaw
  - 145, Warsaw
  - 149, Warsaw
- Spain (6):
  - 187, Alcorcón
  - 181, Barcelona
  - 184, Donostia / San Sebastian
  - 182, Madrid
  - 183, Vigo
  - 185, Zaragoza
- Switzerland (5):
  - 201, Biel
  - 205, Geneva
  - 203, Sankt Gallen
  - 202, Tschugg
  - 204, Zurich
- United Kingdom (2):
  - 223, Liverpool
  - 224, Middlesbrough

REFERENCES:
- [Result] Ryvlin P, Werhahn KJ, Blaszczyk B, Johnson ME, Lu S. Adjunctive brivaracetam in adults with uncontrolled focal epilepsy: results from a double-blind, randomized, placebo-controlled trial. Epilepsia. 2014 Jan;55(1):47-56. doi: 10.1111/epi.12432. Epub 2013 Oct 28. PMID 24256083
- [Result] Toledo M, Whitesides J, Schiemann J, Johnson ME, Eckhardt K, McDonough B, Borghs S, Kwan P. Safety, tolerability, and seizure control during long-term treatment with adjunctive brivaracetam for partial-onset seizures. Epilepsia. 2016 Jul;57(7):1139-51. doi: 10.1111/epi.13416. Epub 2016 Jun 6. PMID 27265725
- [Result] Ben-Menachem E, Mameniskiene R, Quarato PP, Klein P, Gamage J, Schiemann J, Johnson ME, Whitesides J, McDonough B, Eckhardt K. Efficacy and safety of brivaracetam for partial-onset seizures in 3 pooled clinical studies. Neurology. 2016 Jul 19;87(3):314-23. doi: 10.1212/WNL.0000000000002864. Epub 2016 Jun 22. PMID 27335114
- [Result] Brodie MJ, Whitesides J, Schiemann J, D'Souza J, Johnson ME. Tolerability, safety, and efficacy of adjunctive brivaracetam for focal seizures in older patients: A pooled analysis from three phase III studies. Epilepsy Res. 2016 Nov;127:114-118. doi: 10.1016/j.eplepsyres.2016.08.018. Epub 2016 Aug 18. PMID 27589414
- [Result] Mukuria C, Young T, Keetharuth A, Borghs S, Brazier J. Sensitivity and responsiveness of the EQ-5D-3L in patients with uncontrolled focal seizures: an analysis of Phase III trials of adjunctive brivaracetam. Qual Life Res. 2017 Mar;26(3):749-759. doi: 10.1007/s11136-016-1483-3. Epub 2016 Dec 21. PMID 28004320
- [Result] Moseley BD, Sperling MR, Asadi-Pooya AA, Diaz A, Elmouft S, Schiemann J, Whitesides J. Efficacy, safety, and tolerability of adjunctive brivaracetam for secondarily generalized tonic-clonic seizures: Pooled results from three Phase III studies. Epilepsy Res. 2016 Nov;127:179-185. doi: 10.1016/j.eplepsyres.2016.09.003. Epub 2016 Sep 3. PMID 27608437
- [Result] Brandt C, Borghs S, Elmoufti S, Mueller K, Townsend R, de la Loge C. Health-related quality of life in double-blind Phase III studies of brivaracetam as adjunctive therapy of focal seizures: A pooled, post-hoc analysis. Epilepsy Behav. 2017 Apr;69:80-85. doi: 10.1016/j.yebeh.2016.11.031. Epub 2017 Feb 23. PMID 28236727
- [Result] Klein P, Johnson ME, Schiemann J, Whitesides J. Time to onset of sustained >/=50% responder status in patients with focal (partial-onset) seizures in three phase III studies of adjunctive brivaracetam treatment. Epilepsia. 2017 Feb;58(2):e21-e25. doi: 10.1111/epi.13631. Epub 2016 Dec 18. PMID 27988967
- [Result] Asadi-Pooya AA, Sperling MR, Chung S, Klein P, Diaz A, Elmoufti S, Schiemann J, Whitesides J. Efficacy and tolerability of adjunctive brivaracetam in patients with prior antiepileptic drug exposure: A post-hoc study. Epilepsy Res. 2017 Mar;131:70-75. doi: 10.1016/j.eplepsyres.2017.02.007. Epub 2017 Feb 27. PMID 28279891
- [Result] Benbadis S, Klein P, Schiemann J, Diaz A, Elmoufti S, Whitesides J. Efficacy, safety, and tolerability of brivaracetam with concomitant lamotrigine or concomitant topiramate in pooled Phase III randomized, double-blind trials: A post-hoc analysis. Epilepsy Behav. 2018 Mar;80:129-134. doi: 10.1016/j.yebeh.2017.12.024. Epub 2018 Feb 3. PMID 29414542
- [Result] Brodie MJ, Fakhoury T, McDonough B, Colson AO, Stockis A, Elmoufti S, Whitesides J. Brivaracetam-induced elevation of carbamazepine epoxide levels: A post-hoc analysis from the clinical development program. Epilepsy Res. 2018 Sep;145:55-62. doi: 10.1016/j.eplepsyres.2018.06.002. Epub 2018 Jun 4. PMID 29908435
- [Result] Klein P, Laloyaux C, Elmoufti S, Gasalla T, Martin MS. Time course of 75%-100% efficacy response of adjunctive brivaracetam. Acta Neurol Scand. 2020 Aug;142(2):175-180. doi: 10.1111/ane.13287. Epub 2020 Jun 9. PMID 32432339
- [Result] Moseley BD, Dimova S, Elmoufti S, Laloyaux C, Asadi-Pooya AA. Long-term efficacy and tolerability of adjunctive brivaracetam in adults with focal to bilateral tonic-clonic (secondary generalized) seizures: Post hoc pooled analysis. Epilepsy Res. 2021 Oct;176:106694. doi: 10.1016/j.eplepsyres.2021.106694. Epub 2021 Jun 24. PMID 34218211
- [Result] Ryvlin P, Dimova S, Elmoufti S, Floricel F, Laloyaux C, Nondonfaz X, Biton V. Tolerability and efficacy of adjunctive brivaracetam in adults with focal seizures by concomitant antiseizure medication use: Pooled results from three phase 3 trials. Epilepsia. 2022 Aug;63(8):2024-2036. doi: 10.1111/epi.17304. Epub 2022 Jun 10. PMID 35582748
- [Derived] Bresnahan R, Panebianco M, Marson AG. Brivaracetam add-on therapy for drug-resistant epilepsy. Cochrane Database Syst Rev. 2022 Mar 14;3(3):CD011501. doi: 10.1002/14651858.CD011501.pub3. PMID 35285519
- [Derived] Lee SK, Heo K, Kim SE, Lee SA, Elmoufti S, Laloyaux C, Hur B. Effect of Number of Previous Antiseizure Medications on Efficacy and Tolerability of Adjunctive Brivaracetam for Uncontrolled Focal Seizures: Post Hoc Analysis. Adv Ther. 2021 Jul;38(7):4082-4099. doi: 10.1007/s12325-021-01816-5. Epub 2021 Jun 21. PMID 34155568
- [Derived] Ben-Menachem E, Baulac M, Hong SB, Cleveland JM, Reichel C, Schulz AL, Wagener G, Brandt C. Safety, tolerability, and efficacy of brivaracetam as adjunctive therapy in patients with focal seizures, generalized onset seizures, or Unverricht-Lundborg disease: An open-label, long-term follow-up trial. Epilepsy Res. 2021 Feb;170:106526. doi: 10.1016/j.eplepsyres.2020.106526. Epub 2020 Dec 4. PMID 33461041

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study started to enroll subjects in September 2007 and concluded in February 2009.
Pre-assignment Details: Participant Flow refers to the Randomized Set.
Period: Overall Study
Arm/Group | Placebo | Brivaracetam 20 mg/Day | Brivaracetam 50 mg/Day | Brivaracetam 100 mg/Day
Started | 100 | 99 | 100 | 100
Completed | 92 | 93 | 88 | 94
Not Completed | 8 | 6 | 12 | 6
Not completed — AE, non-serious non-fatal | 3 | 4 | 4 | 5
Not completed — Lost to Follow-up | 2 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 0
Not completed — Other reason | 0 | 1 | 3 | 1
Not completed — AE, serious fatal | 1 | 0 | 0 | 0
Not completed — Serious adverse event (SAE), non-fatal | 0 | 0 | 1 | 0
Not completed — AE of unknown type | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Randomized Set.
Arm/Group | Placebo | Brivaracetam 20 mg/Day | Brivaracetam 50 mg/Day | Brivaracetam 100 mg/Day | Total Title
Number analyzed (Participants) | 100 | 99 | 100 | 100 | 399
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.4 (13.0) | 35.7 (12.5) | 39.0 (13.5) | 38.0 (13.1) | 37.24 (13.05)
Age, Customized [Number; unit: participants]
  <18 years | 2 | 2 | 0 | 1 | 5
  Between 18 and 65 years | 96 | 94 | 97 | 96 | 383
  >=65 years | 2 | 3 | 3 | 3 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 38 | 45 | 42 | 171
  Male | 54 | 61 | 55 | 58 | 228
Region of Enrollment [Number; unit: Participants]
  Hungary | 4 | 2 | 3 | 3 | 12
  Poland | 26 | 28 | 27 | 27 | 108
  India | 23 | 22 | 23 | 23 | 91
  Belgium | 3 | 0 | 3 | 0 | 6
  Finland | 3 | 3 | 1 | 4 | 11
  France | 17 | 17 | 11 | 15 | 60
  Germany | 8 | 10 | 14 | 9 | 41
  Italy | 4 | 8 | 3 | 5 | 20
  Netherlands | 3 | 0 | 1 | 3 | 7
  Spain | 8 | 4 | 6 | 4 | 22
  Switzerland | 1 | 3 | 6 | 5 | 15
  United Kingdom | 0 | 2 | 2 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Partial Onset Seizure (Type I) Frequency Per Week Over the 12-week Treatment Period
Description: Partial (Type I) Seizures can be classified into one of the following three groups: Simple Partial Seizures, Complex Partial Seizures, Partial Seizures evolving to Secondarily Generalized Seizures.
Time Frame: From Baseline to 12-week Treatment Period
Population: The Intention-to-treat (ITT) population was defined as all randomized subjects who received at least 1 dose of study medication.
Measure: Median (Inter-Quartile Range); unit: Seizure Frequency per Week
Arm/Group | Placebo | Brivaracetam 20 mg/Day | Brivaracetam 50 mg/Day | Brivaracetam 100 mg/Day
Number analyzed (Participants) | 100 | 99 | 99 | 100
Seizure Frequency per Week | 1.75 [0.76 to 5.12] | 1.34 [0.70 to 3.12] | 1.49 [0.69 to 2.78] | 1.26 [0.52 to 2.93]
Statistical Analysis 1: Comparison: Placebo vs Brivaracetam 50 mg/Day; In order to control the Type I error testing was performed in sequence starting with 50 mg, then 100 mg and finally 20 mg Brivaracetam per day versus Placebo, only moving to the next test if the previous one was significant at the 5 % level; Test type: Superiority or Other; p = 0.261, ANCOVA; Percentage Reduction over Placebo = 6.5, 95% CI 2-sided [-5.2 to 16.9]

2. Secondary Outcome: Responder Rate for Partial Onset Seizures (Type I) Frequency Per Week Over the 12-week Treatment Period
Description: Responders are those subjects with at least 50 % reduction from Baseline to Treatment Period in Partial Onset Seizure frequency per week.
  The Responder Rate for Partial Onset Seizures (Type I) is the proportion of subjects who have a >= 50 % reduction in seizure frequency per week from Baseline.
Time Frame: From Baseline to 12-week Treatment Period
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Brivaracetam 20 mg/Day | Brivaracetam 50 mg/Day | Brivaracetam 100 mg/Day
Number analyzed (Participants) | 100 | 99 | 99 | 100
Percentage of Participants
  Non-responders | 80.0 | 72.7 | 72.7 | 64.0
  Responders | 20.0 | 27.3 | 27.3 | 36.0

3. Secondary Outcome: All Seizure Frequency (Type I+II+III) Per Week Over the 12-week Treatment Period
Description: There are three types of Epilepsy: Partial Epilepsies (Type I), Generalized Epilepsies (Type II) and uncertain classification of Epilepsies (Type III).
Time Frame: From Baseline to 12-week Treatment Period
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Times per week
Arm/Group | Placebo | Brivaracetam 20 mg/Day | Brivaracetam 50 mg/Day | Brivaracetam 100 mg/Day
Number analyzed (Participants) | 100 | 99 | 99 | 100
Times per week | 1.75 [0.76 to 5.61] | 1.34 [0.70 to 3.12] | 1.49 [0.69 to 2.78] | 1.26 [0.52 to 2.93]

4. Secondary Outcome: Percent Change From Baseline to the 12-week Treatment Period in Partial Onset Seizure (Type I) Frequency Per Week
Description: The percent change from Baseline was computed as: Weekly Seizure Frequency (Treatment) - Weekly Seizure Frequency (Baseline) / Weekly Seizure Frequency (Baseline) * 100. Negative values indicate a reduction from Baseline with higher negative values showing higher reduction.
Time Frame: From Baseline to 12-week Treatment Period
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percent change in seizures per week
Arm/Group | Placebo | Brivaracetam 20 mg/Day | Brivaracetam 50 mg/Day | Brivaracetam 100 mg/Day
Number analyzed (Participants) | 100 | 99 | 99 | 100
Percent change in seizures per week | -17.03 [-40.27 to 17.59] | -30.03 [-55.99 to -2.11] | -26.83 [-60.05 to 6.32] | -32.45 [-72.51 to 0.04]

5. Secondary Outcome: Categorized Percentage Change From Baseline in Seizure Frequency for Partial Onset Seizure (Type I) Over the 12-week Treatment Period
Description: The categories are:
  * <= 25 %
  * - 25 % to < 25 %
  * 25 % to < 50 %
  * 50 % to < 75 %
  * 75 % to < 100 %
  * 100 %
Time Frame: From Baseline to 12-week Treatment Period
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Brivaracetam 20 mg/Day | Brivaracetam 50 mg/Day | Brivaracetam 100 mg/Day
Number analyzed (Participants) | 100 | 99 | 99 | 100
Percentage of Participants
  <= 25 % | 19.0 | 10.1 | 15.2 | 10.0
  - 25 % to < 25 % | 41.0 | 35.4 | 33.3 | 33.0
  25 % to < 50 % | 20.0 | 27.3 | 24.2 | 21.0
  50 % to < 75 % | 12.0 | 18.2 | 17.2 | 14.0
  75 % to < 100 % | 8.0 | 7.1 | 9.1 | 18.0
  100 % | 0 | 2.0 | 1.0 | 4.0

6. Secondary Outcome: Seizure Freedom Rate (All Seizure Types) Over the 12-week Treatment Period
Description: Subjects were considered seizure free if their seizure counts for every day over the entire Treatment Period was zero and if they completed the Treatment Period.
Time Frame: From Baseline to 12-week Treatment Period
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Brivaracetam 20 mg/Day | Brivaracetam 50 mg/Day | Brivaracetam 100 mg/Day
Number analyzed (Participants) | 100 | 99 | 99 | 100
Percentage of Participants
  Seizure free | 0 | 2.0 | 0 | 4.0
  No Seizures but non-completer | 0 | 0 | 1.0 | 0
  Not Seizure-free | 100.0 | 98.0 | 99.0 | 96.0

7. Secondary Outcome: Time to First Type I Seizure During the 12-week Treatment Period
Description: The time to first Type I Seizure during the 12-week Treatment Period was measured in days.
Time Frame: From Baseline to 12-week Treatment Period
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | Brivaracetam 20 mg/Day | Brivaracetam 50 mg/Day | Brivaracetam 100 mg/Day
Number analyzed (Participants) | 100 | 99 | 99 | 100
Days | 4 [3 to 5] | 6 [3 to 8] | 6 [4 to 10] | 4 [3 to 5]

8. Secondary Outcome: Time to Fifth Type I Seizure During the 12-week Treatment Period
Description: The time to Fifth Type I Seizure during the 12-week Treatment Period was measured in days.
Time Frame: From Baseline to 12-week Treatment Period
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | Brivaracetam 20 mg/Day | Brivaracetam 50 mg/Day | Brivaracetam 100 mg/Day
Number analyzed (Participants) | 100 | 99 | 99 | 100
Days | 19 [14 to 25] | 25 [20 to 34] | 24 [20 to 32] | 24 [18 to 34]

9. Secondary Outcome: Time to Tenth Type I Seizure During the 12-week Treatment Period
Description: The time to tenth Type I Seizure during the 12-week Treatment Period was measured in days.
Time Frame: From Baseline to 12-week Treatment Period
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | Brivaracetam 20 mg/Day | Brivaracetam 50 mg/Day | Brivaracetam 100 mg/Day
Number analyzed (Participants) | 100 | 99 | 99 | 100
Days | 39 [24 to 50] | 49 [36 to 64] | 40 [33 to 49] | 46 [34 to 66]

10. Secondary Outcome: Reduction of Type IC/Type I Seizure Frequency Ratio From Baseline to the 12- Week Treatment Period.
Description: The type IC/Type I seizure frequency ratio is represented by the percentage of subjects having a reduction in the ratio of Type IC seizure frequency over Type IA, IB, and IC seizure frequency from Baseline to Treatment Period.
Time Frame: From Baseline to 12-week Treatment Period
Population: The Intention-to-treat (ITT) population was defined as all randomized subjects who received at least 1 dose of study medication.
  Type IC Population consists of those subjects with at least one Type IC seizure during the Baseline period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Brivaracetam 20 mg/Day | Brivaracetam 50 mg/Day | Brivaracetam 100 mg/Day
Number analyzed (Participants) | 37 | 36 | 40 | 39
percentage of participants | 45.9 | 47.2 | 62.5 | 41.0

11. Secondary Outcome: Change From Baseline to the 12-week Treatment Period in Total Patient Weighted Quality of Life in Epilepsy Inventory-Form 31 (QOLIE-31-P) Score
Description: The QOLIE-31-P is an adaptation of the original QOLIE-31 instrument that includes 30 items grouped into seven multi-item subscales - Seizure Worry (5 items), Overall Quality of Life (2 items), Emotional Well-Being (5 items), Energy/Fatigue (4 items), Cognitive Functioning (6 items), Medication Effects (3 items) and Daily Activities/Social Functioning (5 items) - and a Health Status item. The subscale scores, the Total score and the Health Status item score are calculated according to the scoring algorithm defined by the author with scores ranging from 0 to 100 and higher scores indicating better function. A positive value in Change from Baseline indicates an improvement from Baseline.
Time Frame: From Baseline to 12-week Treatment Period
Population: Subjects in the Intention-To-Treat (ITT) population with measurements at Baseline and Last Visit / Early Discontinuation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Brivaracetam 20 mg/Day | Brivaracetam 50 mg/Day | Brivaracetam 100 mg/Day
Number analyzed (Participants) | 86 | 91 | 94 | 80
units on a scale | 2.29 (14.03) | 4.50 (12.71) | 3.09 (14.43) | 1.78 (13.95)

12. Secondary Outcome: Change From Baseline to the 12-week Treatment Period in Seizure Worry Patient Weighted Quality of Life in Epilepsy Inventory-Form 31 (QOLIE-31-P) Score
Description: as for outcome 11
Time Frame: From Baseline to 12-week Treatment Period
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Brivaracetam 20 mg/Day | Brivaracetam 50 mg/Day | Brivaracetam 100 mg/Day
Number analyzed (Participants) | 88 | 93 | 96 | 86
units on a scale | 8.25 (22.01) | 6.23 (17.97) | 5.34 (23.81) | 8.04 (26.26)

13. Secondary Outcome: Change From Baseline to the 12-week Treatment Period in Daily Activities/Social Functioning Patient Weighted Quality of Life in Epilepsy Inventory-Form 31 (QOLIE-31-P) Score
Description: as for outcome 11
Time Frame: From Baseline to 12-week Treatment Period
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Brivaracetam 20 mg/Day | Brivaracetam 50 mg/Day | Brivaracetam 100 mg/Day
Number analyzed (Participants) | 88 | 93 | 96 | 85
units on a scale | -2.09 (20.26) | 3.35 (19.72) | 3.09 (20.79) | 3.50 (22.52)

14. Secondary Outcome: Change From Baseline to the 12-week Treatment Period in Hospital Anxiety Score
Description: The Hospital Anxiety and Depression Scale (HADS) was used to evaluate anxiety and depression simultaneously. The HADS was developed as a self-administered scale that has been designed to assess the presence and severity of both anxiety and depression. It consists of 14 items that are scored on a 4-point severity scale ranging from 0 to 3. A score per dimension was calculated with each score ranging from 0 to 21 and higher scores indicating higher depression / anxiety. Negative values in Change from Baseline indicate a decrease of HADS from Baseline to Treatment Period.
Time Frame: From Baseline to 12-week Treatment Period
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Brivaracetam 20 mg/Day | Brivaracetam 50 mg/Day | Brivaracetam 100 mg/Day
Number analyzed (Participants) | 86 | 91 | 95 | 83
units on a scale | -1.54 (3.89) | -0.59 (3.89) | -0.41 (3.82) | 0.08 (3.60)

15. Secondary Outcome: Change From Baseline to the 12-week Treatment Period in Hospital Depression Score
Description: as for outcome 14
Time Frame: From Baseline to 12-week Treatment Period
Population: Subjects in the Intention-to-treat (ITT) population with measurements at Baseline and Last Visit / Early Discontinuation Visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Brivaracetam 20 mg/Day | Brivaracetam 50 mg/Day | Brivaracetam 100 mg/Day
Number analyzed (Participants) | 86 | 91 | 95 | 83
units on a scale | -0.65 (3.58) | -0.10 (3.67) | 0.26 (3.84) | -0.24 (3.69)

16. Secondary Outcome: Patient's Global Evaluation Scale (P-GES) Evaluated at Last Visit or Early Discontinuation Visit
Description: The Patient's Global Evaluation Scale (P-GES) is a global assessment of the disease evolution which was performed using a seven-point scale (1 = Marked worsening to 7 = Marked improvement) with the start of the study medication as the reference time point. The subject not mentally impaired had to complete it by answering the following question: "Overall, has there been a change in your seizures since the start of the study medication?"
Time Frame: Last Visit or Early Discontinuation Visit in the 12-week Treatment Period
Population: Subjects in the Intention-to-treat (ITT) population with measurements at Baseline and Last Visit or Early Discontinuation Visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Brivaracetam 20 mg/Day | Brivaracetam 50 mg/Day | Brivaracetam 100 mg/Day
Number analyzed (Participants) | 81 | 90 | 90 | 85
units on a scale | 4.93 (1.39) | 5.17 (1.27) | 5.04 (1.29) | 5.47 (1.16)

17. Secondary Outcome: Investigator's Global Evaluation Scale (I-GES) Evaluated at Last Visit or Early Discontinuation Visit
Description: The Investigator's Global Evaluation Scale (I-GES) is a global assessment of the disease evolution which was performed using a seven-point scale (1 = Marked worsening to 7 = Marked improvement), with the start of the study medication as reference time point. The Investigator was to complete it by answering the following question: "Assess the Overall change in the severity of patient's illness, compared to start of study medication."
Time Frame: Last Visit or Early Discontinuation Visit in the 12-week Treatment Period
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Brivaracetam 20 mg/Day | Brivaracetam 50 mg/Day | Brivaracetam 100 mg/Day
Number analyzed (Participants) | 96 | 99 | 98 | 100
units on a scale | 4.78 (1.20) | 4.99 (1.15) | 4.99 (1.10) | 5.34 (1.12)

18. Secondary Outcome: Change From Baseline to the 12-week Treatment Period in Energy/Fatigue Patient Weighted Quality of Life in Epilepsy Inventory-Form 31 (QOLIE-31-P) Score
Description: as for outcome 11
Time Frame: From Baseline to 12-week Treatment Period
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Brivaracetam 20 mg/Day | Brivaracetam 50 mg/Day | Brivaracetam 100 mg/Day
Number analyzed (Participants) | 86 | 92 | 95 | 83
units on a scale | 3.49 (19.22) | 3.53 (17.04) | 1.95 (20.74) | 1.99 (20.42)

19. Secondary Outcome: Change From Baseline to the 12-week Treatment Period in Emotional Well-Being Patient Weighted Quality of Life in Epilepsy Inventory-Form 31 (QOLIE-31-P) Score
Description: as for outcome 11
Time Frame: From Baseline to 12-week Treatment Period
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Brivaracetam 20 mg/Day | Brivaracetam 50 mg/Day | Brivaracetam 100 mg/Day
Number analyzed (Participants) | 88 | 93 | 96 | 84
units on a scale | 3.80 (18.71) | 3.75 (15.94) | 3.13 (19.35) | -2.45 (18.55)

20. Secondary Outcome: Change From Baseline to the 12-week Treatment Period in Cognitive Functioning Patient Weighted Quality of Life in Epilepsy Inventory-Form 31 (QOLIE-31-P) Score
Description: as for outcome 11
Time Frame: From Baseline to 12-week Treatment Period
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Brivaracetam 20 mg/Day | Brivaracetam 50 mg/Day | Brivaracetam 100 mg/Day
Number analyzed (Participants) | 88 | 93 | 96 | 85
units on a scale | 1.80 (19.16) | 5.36 (20.69) | 1.02 (19.95) | 0.69 (16.66)

21. Secondary Outcome: Change From Baseline to the 12-week Treatment Period in Medication Effects Patient Weighted Quality of Life in Epilepsy Inventory-Form 31 (QOLIE-31-P) Score
Description: as for outcome 11
Time Frame: From Baseline to 12-week Treatment Period
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Brivaracetam 20 mg/Day | Brivaracetam 50 mg/Day | Brivaracetam 100 mg/Day
Number analyzed (Participants) | 88 | 92 | 96 | 86
units on a scale | 0.92 (28.93) | 3.64 (29.24) | -0.85 (24.36) | 3.00 (28.22)

22. Secondary Outcome: Change From Baseline to the 12-week Treatment Period in Overall Quality of Life Patient Weighted Quality of Life in Epilepsy Inventory-Form 31 (QOLIE-31-P) Score
Description: as for outcome 11
Time Frame: From Baseline to 12-week Treatment Period
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Brivaracetam 20 mg/Day | Brivaracetam 50 mg/Day | Brivaracetam 100 mg/Day
Number analyzed (Participants) | 88 | 93 | 95 | 86
units on a scale | 5.11 (18.48) | 4.52 (16.73) | 4.55 (18.93) | 2.24 (18.45)

23. Secondary Outcome: Change From Baseline to the 12-week Treatment Period in Health Status of Life Patient Weighted Quality of Life in Epilepsy Inventory-Form 31 (QOLIE-31-P) Score
Description: as for outcome 11
Time Frame: From Baseline to 12-week Treatment Period
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Brivaracetam 20 mg/Day | Brivaracetam 50 mg/Day | Brivaracetam 100 mg/Day
Number analyzed (Participants) | 88 | 93 | 95 | 84
units on a scale | 6.6 (16.3) | 6.9 (20.1) | 9.7 (19.8) | 4.9 (18.1)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected up to 23 weeks from Visit 1 (Week -8) to the Safety Visit (Week 15).
Description: Adverse Events (AEs) refer to the Safety Set (SS) population wich contains the same set of subjects as the Intention-To-Treat (ITT) population.
Arm/Group | Placebo | Brivaracetam 20 mg/Day | Brivaracetam 50 mg/Day | Brivaracetam 100 mg/Day
Serious Adverse Events (participants affected / at risk) | 6/100 | 2/99 | 4/99 | 2/100
Other Adverse Events (participants affected / at risk) | 22/100 | 31/99 | 35/99 | 37/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=100) | Brivaracetam 20 mg/Day (N=99) | Brivaracetam 50 mg/Day (N=99) | Brivaracetam 100 mg/Day (N=100)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Amnesia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 3 (4) | 0 (0) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Grand mal convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psychotic Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Status epilepticus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=100) | Brivaracetam 20 mg/Day (N=99) | Brivaracetam 50 mg/Day (N=99) | Brivaracetam 100 mg/Day (N=100)
Convulsion (Nervous system disorders) | 1 (1) | 5 (7) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 5 (11) | 5 (8) | 7 (12) | 5 (5)
Fatigue (General disorders) | 2 (2) | 3 (4) | 4 (5) | 8 (9)
Headache (Nervous system disorders) | 10 (14) | 14 (19) | 18 (31) | 9 (15)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 8 (8) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (4) | 0 (0) | 1 (1) | 6 (7)
Somnolence (Nervous system disorders) | 6 (6) | 8 (10) | 6 (7) | 8 (8)
Vertigo (Ear and labyrinth disorders) | 3 (5) | 1 (2) | 2 (2) | 8 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days